CLINICAL TRIAL: NCT02366182
Title: Does Neck Circumference Help to Predict Difficult Airway in Obstetric Patients?
Status: Completed | Type: Observational
Sponsor: Corniche Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Ch09101401
Record Dates: First submitted 2015-01-18; First posted 2015-02-19 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Difficult; Intubation, in Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Failed intubation and ventilation in obstetrics remains one of the most common causes of death directly related to anesthesia. The reported incidence of failed intubation in obstetrics is 1:300, which is significantly higher than that in the non-obstetric population. A clinical screening test with high sensitivity and specificity for prediction of difficult airway may help reduce morbidity and mortality from general anesthesia. Few studies have identified increased neck circumference as the best single predictor of problematic intubation. However the cutoff point of this test for identifying patients at high risk of difficult intubation is not clear.

The aim of this study is to determine the optimal cutoff point, which validates prediction of difficult ventilation and/or intubation for obstetric patients. Preoperative airway assessment will be done including neck circumference. Intraoperative difficult ventilation and/or intubation will be recorded. Optimal cutoff point of neck circumference will be calculated by Receiver Operating characteristics (ROC) curve.

DETAILED DESCRIPTION:
In this prospective study, patients will be assessed by the anaesthetist preoperatively and asked about their medical history including detailed history of obstructive sleep apnea (OSA) and snoring. Physical examination including weight,height &BMI .

Airway assessment will include:

1. Maximum mouth opening measured as interincisor gap (mm).
2. Sternomental distance measured as the straight distance between the upper border of manubrium sterni and the bony point of the mentum with the head in full extension and the mouth is closed (cm).
3. Hyomental distance measured from just above the hyoid bone to the tip to the anterior-most part of the mentum in both neutral position and with maximum head extension (cm). Hence, hyomental distance ratio (HMDR) will be calculated.
4. Thyromental distance measured as the distance from the thyroid notch to the inner margin of the mental prominence when the head is fully extended (cm).
5. Extended Mallampati Score (EMS) in sitting position with full extension of craniocervical junction with phonation (class I: Entire Uvula is clearly visible; class II: Upper half of the uvula is visible; class III: soft and hard palate clearly visible; and class IV: Only hard palate is visible).
6. Neck Circumference at the level of the thyroid cartilage (cm).
7. Condition of the teeth (Protrusion, loose, missing).
8. Mandibular protrusion test to detect temporomandibular joint mobility measured as ability to move the lower teeth in front of the upper teeth.

Intubation will be considered difficult if the Intubation Difficulty Scale ( IDS) is equal or more than 5 .

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cesarean section under general anesthesia

Exclusion Criteria:

* Patients with upper airway pathology
* Patients with cervical spine abnormality
* Emergency cesarean section
* Known cases of difficult intubation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients scheduled for cesarean section under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Difficult intubation | 5 minutes
  Difficult intubation defined as Intubation difficulty scale (IDS) >5

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad, MD, Principal Investigator — Corniche Hospital; Tarek Ansari, FFARCSI, Principal Investigator — Corniche Hospital; Nanda Shetty, MD, Principal Investigator — Corniche Hospital
Locations (1):
- Corniche Hospital, Abu Dhabi, United Arab Emirates

REFERENCES:
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711